CLINICAL TRIAL: NCT04669769
Title: Retrospective Analysis of Outcomes After Surgery for Deep Infiltrating Endometriosis of the Bowel
Brief Title: Retrospective Analysis of Results of Surgery for Deep Bowel Endometriosis
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Dr. med. Sebastian Daniel Schäfer, Head of Gynecology, University Hospital Muenster
Other Study IDs: Schäfer_Endo_DIE_Bowel_Com
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Endometriosis; Deep Endometriosis; Bowel Endometriosis; Reproductive Issues; Complication
Keywords: endometriosis; deep endometriosis; bowel endometriosis; conception; ART; spontaneous conception; pregnancy rate
MeSH Terms: conditions — Endometriosis | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- shaving: patients with DIE and shaving
  Interventions: Other: interview
- disc resection: patients with DIE and Disc resection
  Interventions: Other: interview
- segmental resection: patients with DIE and segmental resection
  Interventions: Other: interview
- multifocal: patients with multifocal DIE having more than one bowel procedure
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — telephone interview

SUMMARY:
identification of patients operated becaus of bowel endometriosis at the endometriosis center, University Hospital Muenster, Germany, starting 2009, Analysis of Patient history, surgical procedurie, intraoperative complications, postoperative complications, phone call assessing further complications, complaints after surgery, pregnancy, live birth, additional surgery, spontaneous conception, conception by IUI, ART

ELIGIBILITY:
Inclusion Criteria:

* deep Infiltrating endometriosis, surgery with complete or partial resection of bowel endometriosis or conservative Management, Treatment at endometriosis Center University Hospital Muenster, Germany, wants to participate

Exclusion Criteria:

* declines participation

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: patients treated because of deep Infiltrating bowel endometriosis at the endometriosis Center, University Hospital Muenster, Germany starting 2009
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
complications | up to 10 years
  complications according to Clavien Dindo Classification

SECONDARY OUTCOMES:
pregnancy rate | up to 10 years
  pregancy after surgery
live birth | up to 10 years
  live birth after surgery
pain recurrence | up to 10 years
  pain recurrence after operation
disease recurrence | up to 10 years
  disease recurrence after operation
recurrent surgery | up to 10 years
  recurrent surgery after surgery for bowel endometriosis
pregnancy rate with ongoing bowel endometriosis | up to 10 years
  pregnancy rate with ongoing bowel endometriosis
live birth with ongoing bowel endometriosis | up to 10 years
  live birth with ongoing bowel endometriosis

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian D Schaefer, MD PhD, Principal Investigator — University Hospital Muenster, Germany
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
will be shared upon reasonable request and according to regulations